CLINICAL TRIAL: NCT02129881
Title: The ONE Study: A Unified Approach to Evaluating Cellular Immunotherapy in Solid Organ Transplantation
Brief Title: The ONE Study UK Treg Trial
Acronym: ONETreg1
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Collaborators: King's College London (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ONETreg1
Record Dates: First submitted 2014-05-01; First posted 2014-05-02 (Estimated); Last update posted 2019-01-25 (Actual); Status verified 2019-01

CONDITIONS: End-stage Renal Failure
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Autologous regulatory T Cell Product (Experimental): Autologous regulatory T Cell Product (1-10 million cells/kg) infused intravenously 5 days post renal transplantation. Recipients also receive prednisolone, mycophenolate mofetil, and tacrolimus as detailed below:
  Prednisolone Day 0: 500 mg IV (250mg pre-op, 250mg intra-op) Day 1: 125 mg IV Day 2 to 14: 20.0 mg/day oral Week 3 to 4: 15.0 mg/day oral Week 5 to 8: 10.0 mg/day oral Week 9 to 12: 5.0 mg/day oral Week 13 to 14: 2.5 mg/day oral Week 15 to End: Cessation Mycophenolate Mofetil (MMF) Day -7 to -2: 500 mg/day oral Day -1 to 14: 2000 mg/day oral Week 3 to 36: 1000 mg/day oral Week 37 to 40: 750 mg/day oral Week 41 to 44: 500 mg/day oral Week 45 to 48: 250 mg/day oral Week 49 to End: Cessation Tacrolimus Day -4 to 14: 3-12 ng/ml oral Week 3 to 12: 3-10 ng/ml oral Week 13 to 36: 3-8 ng/ml oral Week 37 to End: 3-6 ng/ml oral
  Interventions: Biological: Autologous regulatory T Cell Product

INTERVENTIONS:
Biological: Autologous regulatory T Cell Product — Autologous regulatory T Cell Product (1-10 million cells/kg) infused intravenously 5 days post renal transplantation. Recipients also receive prednisolone, mycophenolate mofetil, and tacrolimus as detailed in the arm description.

SUMMARY:
A study to assess cell therapy as a treatment to prevent kidney transplant rejection. The trial will involve purification of naturally occurring regulatory T cells (nTregs) from living-donor renal transplant recipients. The cells will then be grown in the laboratory and re-infused into the patient five days after the kidney transplant. This trial is part of an international European Union funded consortium aimed at evaluating cellular immunotherapy in solid organ transplantation (The ONE Study). It is anticipated that immune regulation induced by nTreg therapy can eventually be used to recude the need for conventional immunosuppression in transplant recipients.

DETAILED DESCRIPTION:
Decades of immunosuppressive drug development has produced an array of powerful pharmacological agents, but the various drawbacks with these treatments leaves considerable room for improvement. By harnessing the power of suppressive mechanisms in the human immune system, regulatory cell therapy may be able to support peripheral tolerance and induce a level of donor-specific unresponsiveness that allows for a reduction in the use of conventional immunosuppression in organ transplant recipients. Several alternative regulatory cell types have been identified as potential adjunct immunotherapies for solid organ transplantation and are now approaching a stage of development that would allow clinical testing in an early-stage trial. The EU-funded international ONE study consortium aims to answer the question as to whether Treg treatment, or other immunoregulatory cell-based therapies, can be advanced in the clinical management of solid organ transplant recipients. This particular Treg trial aims to explored the potential of Treg therapy as an adjunct immunosuppressive treatment in living-donor renal transplant recipients through a clinical protocol design shared by other investigators in the ONE study group testing additional regulatory cell therapies in seperate trials.

ELIGIBILITY:
Recipient Inclusion Criteria

1. Chronic renal insufficiency necessitating kidney transplantation and approved to receive a primary kidney allograft from a living donor
2. Aged at least 18 years
3. Able to commence the immunosuppressive regimen at the protocol-specified time point
4. Willing and able to participate in The ONE Study IM and HEC subprojects
5. Signed and dated written informed consent

Exclusion Criteria

1. Patient has previously received any tissue or organ transplant
2. Known contraindication to the protocol-specified treatments / medications
3. Genetically identical to the prospective organ donor at the HLA loci (0-0-0 mismatch)
4. PRA grade > 40% within 6 months prior to enrolment
5. Previous treatment with any desensitisation procedure (with or without IVIg)
6. Concomitant malignancy or history of malignancy within 5 years prior to planned study entry (excluding successfully-treated non-metastatic basal/squamous cell carcinoma of the skin)
7. Evidence of significant local or systemic infection
8. EBV-negative; serologically positive for anti-HIV-1,2; HBsAg; Anti-HBc; Anti-HCV-ab; Anti-HTLV-1,2 or syphilis (Treponema palladium)
9. Significant liver disease, defined as persistently elevated AST and/or ALT levels > 2 x ULN (Upper Limit of Normal range)
10. Malignant or pre-malignant haematological conditions
11. Any uncontrolled medical condition or concurrent disease that could interfere with the study objectives
12. Any condition which, in the judgement of the Investigator, would place the subject at undue risk
13. Ongoing treatment with systemic immunosuppressive drugs at study entry
14. Participation in another clinical trial during the study or within 28 days prior to planned study entry
15. Female patients of child-bearing potential with a positive pregnancy test at enrolment
16. Female patients who are breast-feeding
17. All female patients of child-bearing potential UNLESS:

    1. The patient is willing to maintain a highly effective method of birth control for the duration of the study
    2. The career, lifestyle, or sexual orientation of the patient ensures that there is no risk of pregnancy for the duration of the study (at the discretion of the Investigator)
18. Psychological, familial, sociological or geographical factors potentially hampering compliance with the study protocol and follow-up visit schedule
19. Any form of substance abuse, psychiatric disorder, or other condition that, in the opinion of the Investigator, may invalidate communication with the Investigator and/or designated study personnel
20. Patients unable to freely give their informed consent (e.g. individuals under legal guardianship).

Donor Inclusion Criteria

1. Eligible for live kidney donation
2. Aged at least 18 years
3. An ABO blood type compatible with the organ recipient
4. Willing and able to provide a blood sample for The ONE Study IM Subproject
5. Willing to provide personal and medical/biological data for the trial analysis
6. Signed and dated written informed consent. Exclusion Criteria

1. Genetically identical to the prospective organ recipient at the HLA loci (0-0-0 mismatch) 2. Exposure to any investigational agents at the time of kidney donation, or within 28 days prior to kidney donation 3. Any form of substance abuse, psychiatric disorder, or other condition that, in the opinion of the Investigator, may invalidate communication with the Investigator designated study personnel 4. Subjects unable to freely give their informed consent (e.g. individuals under legal guardianship)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2014-04 (Actual); Primary Completion 2017-03-23 (Actual); Study Completion 2017-03-23 (Actual)

PRIMARY OUTCOMES:
Incidence of biopsy-confirmed acute rejection. | 60 weeks

SECONDARY OUTCOMES:
Time to first acute rejection episode | 60 weeks
Severity of acute rejection episodes | 60 weeks
Total immunosuppressive burden | 60 weeks
Incidence of chronic graft dysfunction | 60 weeks
Incidence of graft loss through rejection | 60 weeks
Incidence of adverse drug reactions | 60 weeks
Incidence of major and/or opportunistic infections | 60 weeks
Incidence of neoplasia. | 60 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Giovanna Lombardi, PhD, Study Director — King's College Hospital NHS Trust
Locations (2):
- United Kingdom (2):
  - Guy's Hospital, London
  - The Oxford Transplant Centre - Churchill Hospital, Oxford

REFERENCES:
- [Derived] McCallion O, Cross AR, Brook MO, Hennessy C, Ferreira R, Trzupek D, Mulley WR, Kumar S, Soares M, Roberts IS, Friend PJ, Lombardi G, Wood KJ, Harden PN, Hester J, Issa F. Regulatory T cell therapy is associated with distinct immune regulatory lymphocytic infiltrates in kidney transplants. Med. 2025 May 9;6(5):100561. doi: 10.1016/j.medj.2024.11.014. Epub 2024 Dec 27. PMID 39731908
- [Derived] Sawitzki B, Harden PN, Reinke P, Moreau A, Hutchinson JA, Game DS, Tang Q, Guinan EC, Battaglia M, Burlingham WJ, Roberts ISD, Streitz M, Josien R, Boger CA, Scotta C, Markmann JF, Hester JL, Juerchott K, Braudeau C, James B, Contreras-Ruiz L, van der Net JB, Bergler T, Caldara R, Petchey W, Edinger M, Dupas N, Kapinsky M, Mutzbauer I, Otto NM, Ollinger R, Hernandez-Fuentes MP, Issa F, Ahrens N, Meyenberg C, Karitzky S, Kunzendorf U, Knechtle SJ, Grinyo J, Morris PJ, Brent L, Bushell A, Turka LA, Bluestone JA, Lechler RI, Schlitt HJ, Cuturi MC, Schlickeiser S, Friend PJ, Miloud T, Scheffold A, Secchi A, Crisalli K, Kang SM, Hilton R, Banas B, Blancho G, Volk HD, Lombardi G, Wood KJ, Geissler EK. Regulatory cell therapy in kidney transplantation (The ONE Study): a harmonised design and analysis of seven non-randomised, single-arm, phase 1/2A trials. Lancet. 2020 May 23;395(10237):1627-1639. doi: 10.1016/S0140-6736(20)30167-7. PMID 32446407
- See also: One Study — http://www.onestudy.org